CLINICAL TRIAL: NCT05287633
Title: Proton Pump Inhibitors Effects on Dyspepsia During Ramadan Fasting
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PPI
Record Dates: First submitted 2020-09-10; First posted 2022-03-18 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Dyspepsia
Keywords: fasting; Proton Pump Inhibitors; dyspepsia
MeSH Terms: conditions — Dyspepsia; Fasting | interventions — Esomeprazole

STUDY DESIGN:
Intervention Model Description: the objective is to evaluate the interest of proton pump inhibitors in subjects with or without GI symptoms who intend to observe fasting in Ramadan. We will compare the effectiveness of proton pump inhibitors to prevent or reduce the signs of dyspepsia during at least Ramadan as compared to placebo.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A : Proton Pump Inhibitors (Active Comparator): Patients are given proton pump inhibitors tablets once a day
  Interventions: Drug: Esomeprazole
- B: Placebo (Placebo Comparator): Patients are given a placebo instead of proton pump inhibitors active drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esomeprazole — Patients are given a box of capsules of which they take 1capsule/day during the month of ramadan
  Other Names: Nexium
  Arms: A : Proton Pump Inhibitors
Drug: Placebo — Patients are given a box of capsules of which they take 1capsule/day during the month of ramadan
  Arms: B: Placebo

SUMMARY:
evaluate the interest of proton pump inhibitors in subjects with or with GI symptoms who intend to observe fasting in Ramadan. The investigators will compare the effectiveness of proton pump inhibitors to prevent or reduce the signs of dyspepsia during Ramadan compared to placebo.

DETAILED DESCRIPTION:
evaluate the interest of proton pump inhibitors in subjects with or with GI symptoms who intend to observe fasting in Ramadan. Investigators will compare the effectiveness of proton pump inhibitors to prevent or reduce the signs of dyspepsia during at least Ramadan compared to placebo.

The study will be conducted at least from April 2019 to at least June 2030.The study is prospective, two parallel groups, randomized controlled and double blind.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Diagnosed GastroDuodenal Ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Overall symptom relief during the 4 weeks of treatment | 30 days after inclusion
  Relief of dyspepsia symptoms during the treatment period according to the decrease of SF-LDQ score

SECONDARY OUTCOMES:
number of days without dyspepsia | 30 days after inclusion
  the number of days with SF-LDQ score <1
quality of life assessment | 30 days after inclusion
  quality of life assessment ccording to the SF-36 score
Patients satisfaction of the treatment | 30 days after inclusion
  Patients satisfaction according to Likert score

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, Professor, Principal Investigator — University of Monastir
Locations (1):
- Emergency department of university hospital Fattouma Bourguiba of Monastir Monastir, Monastir Tunisia, Monastir, Tunisia

REFERENCES:
- [Derived] Hadrich S, Lamti F, Trabelsi I, Dhaoui R, Ben Abdewahed M, Sekma A, Neffati F, Boukadida L, Yaakoubi H, Jaballah R, Bakir A, Youssef R, Zorgati A, Bel Haj Ali K, Beltaief K, Dridi Z, Ben Hamda K, Jomaa W, Chamtouri I, Bendaya Y, Bouchoucha M, Ben Hafaeidh S, Razgallah R, Bouida W, Grissa MH, Sriha A, Khedher S, Khochtali I, Sakly N, Ben Soltane H, Hassine M, Boubaker H, Boukef R, Msolli MA, Nouira S. Randomized trial of the effect of esomeprazole on functional dyspepsia during Ramadan fasting. Sci Rep. 2025 Oct 21;15(1):36535. doi: 10.1038/s41598-025-17532-x. PMID 41120363